CLINICAL TRIAL: NCT02889939
Title: The Impact of High-intensity, Task Specific Training Combined With Environmental Enrichment for Individuals in a Late Phase After Stroke
Brief Title: High-intensity Training in an Enriched Environment in Late Phase After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Wallström och Sjöbloms stiftelse (Unknown); Peter Erikssons minnesfond (Unknown); Back to Life (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EEHITStroke
Record Dates: First submitted 2016-08-23; First posted 2016-09-07 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Stroke; Brain Diseases
Keywords: rehabilitation; recovery of function; environment
MeSH Terms: conditions — Stroke; Brain Diseases

STUDY DESIGN:
Intervention Model Description: A within-subject, repeated-measures design with pretest-posttest evaluation was utilised to assess outcomes after ETT. The intervention was preceded by a baseline period of usual care (UC) for 3 weeks, which also served as a control
Oversight: Data Monitoring Committee: No

ARMS (1):
- UC + ETT (Other): An enriched comprehensive task-specific therapy (ETT) program combining intensive and task-specific therapy with the sensory-motor, social, and cognitive stimulation inherent to environmental enrichment.
  The intervention was preceded by a baseline period of usual care (UC) for 3 weeks, which also served as a control.
  Interventions: Other: UC + ETT

INTERVENTIONS:
Other: UC + ETT — UC: A 3-week UC period, where the participants were not offered any new rehabilitation activities but were allowed to continue their regular treatment for a maximum of 3 hours per week.
  ETT: The rehabilitation facilities were located in a climate that allowed and encouraged both indoor and outdoor activities. The ETT was individually tailored. Participants exercised in the same room/place as the other participants in groups of 4-9. Physical exercise was scheduled 3.5-6 hours per day, 5½ days per week for 3 weeks. The training was characterized by repetitive mass practice of gradually increasing difficulty and noncompensatory strategies, such as enforcing use of the affected side.
  Beyond scheduled activities, participants were encouraged to physically engage themselves in a challenging outdoor environment.

SUMMARY:
We designed an explorative clinical study to assess the effectiveness of an enriched intense and task-oriented therapy program in enhancing motor recovery in patients with moderate to moderately severe hemiplegia after stroke. This enriched comprehensive task-specific therapy (ETT) program combines intensive and task-specific therapy with the sensory-motor, social, and cognitive stimulation inherent to environmental enrichment. We also investigated whether ETT improves gait, balance, upper and lower limb function, and confidence in task performance, health-related quality of life (HRQoL) and reduces fatigue and depression.

DETAILED DESCRIPTION:
Background The brain has a limited ability for repair. However, in recent years it became evident that a remarkable, yet restricted ability for regeneration of neuronal connections exists, with positive implications for the rehabilitation of individuals with stroke. Several studies have shown that stroke-lesioned animals, which are exposed to a so called enriched environment (large cages, group housing of animals, equipped with toys and with possibilities for physical activity and social interactions) show signs of tissue regeneration/plasticity in the brain. Research has shown that rats exposed to this enriched environment are recovering significantly faster from stroke than rats in standard cages, despite the fact that the total tissue loss between the rats did not differ.

Recovery and improvement of motor functions and skills after stroke depend on spontaneous repair processes but also on the reorganization of neural mechanisms by stimuli and demands that are placed on the motor control system. In spite of numerous research studies showing that functional recovery after stroke is possible even many years after the stroke onset, it is unusual for stroke victims to be offered any kind of rehabilitation during later stages.

The combination of modalities in multimodal interventions is thus expected to have a synergistic effect on neuroplasticity in rehabilitation after stroke in humans. In a recent clinical trial, multimodal interventions based on rhythm and music or therapeutic horseback riding improved recovery in the late phase after stroke Nevertheless, novel combinational treatment approaches are needed to promote neuroplasticity and motor recovery after stroke. A priority is to translate promising basic research to clinical settings and to evaluate enriched combinational therapy programs that appear to be more effective than single interventions

A. What is the impact of high intensity task specific goal-directed training combined with environmental enrichment for individuals in a late phase of stroke? B. What are the subjects' experiences of the rehabilitation program? C. What are the biomarkers of successful stroke recovery? D. How does the intervention effect the subjects' walking ability on a detailed level? The study is a within-subject, repeated-measures design with pretest-posttest study, to assess outcomes after ETT. The intervention was preceded by a baseline period of usual care (UC) for 3 weeks, which also served as a control. The trial enrolled Swedish or Norwegian stroke survivors who had applied to a Swedish rehabilitation agency that provides rehabilitation services in Spain.

The physical evaluation was performed in Sweden prior to and after the intervention and 6 months after completion of the intervention / control period. In addition, a three-month follow-up in form of questionnaires was performed.

The outcome measures were:

Modified Motor Assessment Scale according to Uppsala University Hospital (M-MAS UAS) (measuring motor function), measures of walking ability, speed and endurance, dynamic and static balance, fine motor speed and dexterity in the upper limb, motor speed and gross manual dexterity, hand strength, satisfaction with life as a whole, perceived confidence in task performance, health-related quality of life and degree of depression.

Focus group interviews and individual interviews will be conducted with a subgroup of the participants (non aphasic participants) and the statements will be analyzed qualitative using content analyses as the method.

Blood samples will be taken for the analysis of biomarkers, growth factors and inflammatory markers.

Advanced analyses of gait patterns and components will be performed in a motor laboratory, including a subgroup of the participants.

In rehabilitation medicine, the general belief has been that treatment of individuals in the late phase of stroke has no functional impact. The present research program will test against this hypothesis into a clinical trial for patients at more than 6 months after stroke. The biochemical analysis of blood samples and additional preclinical studies will directly to the knowledge about possibilities to enhance brain plasticity also in later phases of stroke. The research will contribute to strengthening the evidence for a promising rehabilitation approach combining elements of focused high-intensity training with environmental enrichment for which there are strong empirical support.

ELIGIBILITY:
Inclusion criteria:

* At least six months and maximum 10 years after the onset of stroke
* Disability grade between 2 and 4 on the Modified Rankin Scale.
* Some degree of hemiparesis, according to the primary outcome measure M-MAS UAS -99, at baseline.
* Approved by the referring / prescribing physician for intensive training
* Medically stable considering cardiovascular conditions
* Cognitive and speech ability that enables instruction, intervention and evaluation
* Ability and willingness to travel to the place of evaluation
* Able to perform sitting transfers independently or with manual assistance

Exclusion criteria:

* Exercise-induced epilepsy.
* Injury, illness or addiction, making the individual unsuitable for participation.
* Having participated in an intense comprehensive rehabilitation program (additional to post-stroke acute- and subacute rehabilitation) at some point within the past six months.
* Scheduled for other treatment with focus on intensive training during the study.
* Use of assistive technology for sitting transfers

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in Modified Motor Assessment Scale score according to Uppsala from baseline to after intervention/control and from baseline to 6 months follow up. | baseline, 3 weeks, 6 months
  Motor function

SECONDARY OUTCOMES:
Change in Six minute walking test from baseline to after intervention/control and from baseline to 6 months follow up. | baseline, 3 weeks, 6 months
  walking endurance
Change in 10 m walk test from baseline to after intervention/control and from baseline to 6 months follow up. | baseline, 3 weeks, 6 months
  walking ability
Change in Box and Blocks test from baseline to after intervention/control and from baseline to 6 months follow up. | baseline, 3 weeks, 6 months
  gross motor speed
Change in JAMAR from baseline to after intervention/control and from baseline to 6 months follow up. | baseline, 3 weeks, 6 months
  grip strength
Change in Nine Hole Peg Test from baseline to after intervention/control and from baseline to 6 months follow up. | baseline, 3 weeks, 6 months
  fine motor speed
Change in Bergs balance scale from baseline to after intervention/control and from baseline to 6 months follow up. | baseline, 3 weeks, 6 months
  balance ability
Change in Life satisfaction checklist from baseline to after intervention/control, from baseline to 3 months follow up and from baseline to 6 months follow up. | baseline, 3 weeks, 3 months, 6 months
  satisfaction with life
Change in Fatigue impact scale from baseline to after intervention/control, from baseline to 3 months follow up and from baseline to 6 months follow up. | baseline, 3 weeks, 3 months, 6 months
  effect of fatigue in daily activities
Change in Falls Efficacy scale from baseline to after intervention/control, from baseline to 3 months follow up and from baseline to 6 months follow up. | baseline, 3 weeks, 3 months, 6 months
  Perceived confidence in task performance
Change in EuroQual 5D from baseline to after intervention/control, from baseline to 3 months follow up and from baseline to 6 months follow up. | baseline, 3 weeks, 3 months, 6 months
  health related quality of life
Change in Montgomery Åsberg depression rating scale from baseline to after intervention/control, from baseline to 3 months follow up and from baseline to 6 months follow up. | baseline, 3 weeks, 3 months, 6 months
  degree of depression
Change in Life situation among spouses after the stroke event questionnaire from baseline to after intervention/control, from baseline to 3 months follow up and from baseline to 6 months follow up. | baseline, 3 weeks, 3 months, 6 months
  life situation among stroke spouses
Change in levels of biomarkers in blood from baseline to after control/intervention and from baseline to 6 months after intervention. | baseline, 3 weeks, 6 months
  Blood samples will be taken for the analysis of biomarkers, growth factors and inflammatory markers.

CONTACTS AND LOCATIONS:
Overall Officials: Lina Bunketorp Käll, PT, PhD, Study Chair — Göteborg University; Georg Kuhn, Professor, Study Chair — Göteborg University; Jean-Luc Af Geijerstam, MD, PhD, Study Chair — Karolinska Institutet
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vive S, Af Geijerstam JL, Kuhn HG, Bunketorp-Kall L. Enriched, Task-Specific Therapy in the Chronic Phase After Stroke: An Exploratory Study. J Neurol Phys Ther. 2020 Apr;44(2):145-155. doi: 10.1097/NPT.0000000000000309. PMID 32118616